CLINICAL TRIAL: NCT06067477
Title: Estimation of the Dietary Requirement for Vitamin D in Ethnic Groups: a Double-blind, Randomised, Dose-response Trial
Brief Title: Estimation of the Dietary Requirement for Vitamin D in Ethnic Groups
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Surrey (Other)
Collaborators: University of Reading (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FHMS 22-23 194 EGA
Record Dates: First submitted 2023-09-20; First posted 2023-10-05 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Vitamin D Deficiency; Immune Health; Muscle Function
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Intervention Model Description: Recruited participants will be randomised to take 400,1000, or 2000 IU for 12 weeks.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vitamin D Supplement 400 IU (Active Comparator): 400 IU (10 µg) of Vitamin D3
  Interventions: Dietary Supplement: Vitamin D Supplement
- Vitamin D Supplement 1000 IU (Active Comparator): 1000 IU (25 µg) of Vitamin D3
  Interventions: Dietary Supplement: Vitamin D Supplement
- Vitamin D Supplement 2000 IU (Active Comparator): 2000 IU (50 µg) of Vitamin D3
  Interventions: Dietary Supplement: Vitamin D Supplement

INTERVENTIONS:
Dietary Supplement: Vitamin D Supplement — Vitamin D Supplement

SUMMARY:
The aim of this study is to perform a double-blind, randomised, dose-response trial of vitamin D3 supplementation in United Kingdom (UK)-dwelling adults of white European, South Asian, and black African/Caribbean ethnicity to investigate the distribution of dietary intakes needed to maintain adequate vitamin D status in winter, as indicated by serum 25(OH)D concentrations at ranges of >25 to 50 nmol/L. In addition, this study will investigate the effect of vitamin D3 supplementation on immune health, muscular strength, and overall health.

DETAILED DESCRIPTION:
The aim of this study is to perform a double-blind, randomised, dose-response trial of vitamin D3 supplementation in United Kingdom (UK)-dwelling adults of white European, South Asian, and black African/Caribbean ethnicity to investigate the distribution of dietary intakes needed to maintain adequate vitamin D status in winter, as indicated by serum 25(OH)D concentrations at ranges of >25 to 50 nmol/L. In addition, this study will investigate the effect of vitamin D3 supplementation on immune health, muscular strength, and overall health. Recruited participants will be randomised to take 400, 1000, or 2000 IU for 12 weeks. Fasting blood samples collected at baseline and 12 weeks will measure biochemical markers of vitamin D status (serum 25(OH)D, calcium, parathyroid hormone, albumin), lipid profile, ferritin, micronutrient status, and immune and inflammatory biomarkers. Muscular strength will be measured using sit-to-stand and grip strength tests. Questionnaires, food diaries, and dosimeters will be used to gather data on lifestyle, physical activity, dietary intake, and sun exposure.

ELIGIBILITY:
Inclusion Criteria:

* British white European, black African/Caribbean, or South Asian (self-reported)
* Living in England for >2 months
* Aged >18 years
* No significant health issues
* English or Urdu speaker

Exclusion Criteria:

* Medical condition or history which might impact study measurements (e.g., ischaemic heart disease, type 1 and type 2 diabetes, thyroid disease, osteoporosis, haematological disease, malignancy)
* Medications known to affect vitamin D metabolism (i.e., hormone replacement therapy, anti-oestrogens treatment, antiepileptic drugs, and breast cancer treatment)
* Pregnant or planning pregnancy during the study period
* Regular use of sun beds
* Having a sun holiday one month prior to commencing study or plans for a sun holiday within the study period. A sun holiday is generally defined as a holiday in a sunny resort outside of the UK. The researchers will assess this on a case-by-case basis depending on the time of year and expected weather conditions
* Reported participation in another clinical trial occurring simultaneously
* Previous intolerance or allergic reaction to vitamin D

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Concentration of serum 25(OH)D (nmol/L) | Baseline and 12 weeks
  A blood sample will be analysed using liquid chromatography tandem mass spectroscopy (LC-MS). Dose-response change in serum 25(OH)D will be measured in nmol/L.

SECONDARY OUTCOMES:
Anthropometric measurements - weight (kg) | Baseline and 12 weeks
  Weight (kg)
Anthropometric measurements - height (m) | Baseline and 12 weeks
  Height (m)
Anthropometric measurements - height (cm) | Baseline and 12 weeks
  Height (cm)
Anthropometric measurements - waist circumference (cm) | Baseline and 12 weeks
  Waist circumference measurement (cm)
Anthropometric measurements - hip circumference (cm) | Baseline and 12 weeks
  Hip circumference measurement (cm)
Concentration of serum calcium (nmol/L) | Baseline and 12 weeks
  Measure dose-response change in serum calcium measured in nmol/L
Concentration of plasma parathyroid hormone (PTH) (pg/mL) | Baseline and 12 weeks
  Measure dose-response change in plasma parathyroid hormone (PTH) measured in pg/mL
Concentration of serum albumin (g/L) | Baseline and 12 weeks
  Measure dose-response change in serum albumin measured in g/L
Concentration of C-Reactive Protein (CRP) (mg/L) | Baseline and 12 weeks
  Measure dose-response change in CRP measured in mg/L
Complete blood count | Baseline and 12 weeks
  Measure change in complete blood count
Change in immune parameters | Baseline and 12 weeks
  Measure change in gene expression in white blood cells
Number of participants with Acute Respiratory Tract Infections (ARTIs) | 12 weeks
  Measure the frequency of ARTIs using a validated questionnaire
Muscular strength using a handgrip strength test (kg) | Baseline and 12 weeks
  Muscular strength measured using a dynamometer (measured to the nearest 0.1kg). The participant will squeeze the dynamometer with maximum effort for 5 seconds.
Muscular strength and endurance using a sit-to-stand test | Baseline and 12 weeks
  Number of sit to stands in 30 seconds
Blood analytes - micronutrient status | Baseline and 12 weeks
  Measure dose-response change in micronutrient status from blood samples
Blood analytes - lipid profile (mg/dL) | Baseline and 12 weeks
  Measure change in lipid profile from blood samples measured in mg/dL
Vitamin D consumption from diet | Baseline and 12 weeks
  Vitamin D intake will be measured through a 4-day food diary which participants will fill out for 4 day at home before and after the study.
Physical activity questionnaire | Baseline
  Assess level of physical activity using an International Physical Activity Questionnaire (short form)
Sun exposure behaviour questionnaire | Baseline
  Measures amount of time spent in the sun (often, occasionally, never) and what parts of the body are exposed (head, hands, arms, legs, torso) over summer, spring, autumn and winter. Also questions any summer holidays abroad, in what month, what country was visited, number of hours of sun per day and what body parts were exposed (head, hands, arms, legs, torso)
Ultraviolet B radiation (UVB) sun exposure | Baseline and 12 weeks
  Sun exposure will be measured by a dosimeter, which measures UVB exposure. Participants wear this like a badge for 4 days before and after the study.
Lifestyle questionnaire | Baseline
  Measures:
  - Skin type (Fitzpatrick scale)
  Questions:
  Questions what ethnicity they identify with, Holidays abroad, Education, Origin, Health, Pregnancy, Sun behaviours (what body parts are usually exposed to the sun, clothing, sun bathing, sunscreen use, sun bed use), Smoking, Drinking, Recreational drug use, Knowledge around vitamin D, supplement use, Milk, egg, oily fish and liver consumption

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Bournot, Principal Investigator — University of Surrey
Locations (1):
- Faculty of Health and Medical Sciences, Guildford, United Kingdom

IPD SHARING:
Plan to Share IPD: No